CLINICAL TRIAL: NCT04707885
Title: Clinical Utility of Residual Hearing in the Cochlear Implant Ear
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Oliver Adunka, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020H0477; U01DC018920-01 (NIH)
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss; Hearing Loss, Bilateral
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss; Hearing Loss, Bilateral | interventions — Audiometry, Evoked Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ECochG monitoring (Experimental): For those randomized to the experimental group, the CI surgery will proceed in a standard fashion. However, the surgeon will utilize ECochG-guided monitoring by placing the external device coil and processor over the receiver/stimulator of the implanted components. Also, a sound applicator (i.e. speaker) will be placed in the external auditory canal by the surgeon. During electrode insertion the surgeon will utilize the ECochG feedback to adjust insertion if needed. That is, once the electrode has been inserted at least 75% (75% of the electrode contacts inside the cochlea), the surgeon may proceed to full insertion if indicated during ECochG feedback or may modify and/or cease electrode insertion if indicated by the ECochG feedback in attempts to preserve RH.
  Interventions: Device: Electrocochleography
- Control Group (No Intervention): For those randomized to the control group, they will receive their CI per the standard of care. That is, all procedures that take place during a routine CI surgery will be the same for those in the control group. As such, no ECochG monitoring will be performed. However, all study surgeons will be asked to adhere to soft surgical principles (non-traumatic cochlear opening, slow electrode insertions) to enhance HP outcomes even in the absence of intraoperative ECochG monitoring. Further, the standard of care for cochlear implantation is to perform full electrode insertions with all electrode contacts inside of the cochlea. Thus, for subjects in the control group, surgeons will be asked to perform full electrode insertions.

INTERVENTIONS:
Device: Electrocochleography — The use of ECochG monitoring will be employed. This will be conducted intraoperatively during the entire portion of the CI electrode insertion component.
  For the purposes of this clinical trial, the stimulus will consist of a 500 Hz tone burst presented at ~105-110 dB SPL. This was chosen due to the time and resource limitations in the operating room. Hence, the surgical team can only utilize a very limited dataset for intraoperative decision making and previous studies have demonstrated that 500 Hz stimulation offers the most robust, reliable, and useful ECochG signal during electrode insertions.
  Other Names: ECochG
  Arms: ECochG monitoring

SUMMARY:
The current study is a randomized multi-center clinical trial that investigates the role an intraoperative hearing monitoring system (electrocochleography) has on helping to save residual hearing in patients undergoing cochlear implantation (CI).

DETAILED DESCRIPTION:
The clinical importance of residual acoustic hearing in CI remains unclear. It is estimated that only five percent of adult candidates undergo CI. A major barrier is the loss of residual hearing associated with surgery, meaning most patients lose any or all residual hearing as a result of the CI surgery, especially since the majority of today's candidates do not suffer from complete deafness. Hence, many candidates are faced with the decision to relinquish their remaining acoustic hearing in exchange for electric hearing via the CI, as CI surgery often results in complete loss of any residual hearing. However, recent developments in hearing monitoring systems during CI surgery have shown promise for providing the surgeon with live feedback of how the cochlear implant insertion process is proceeding, allowing the surgeon to make intraoperative adjustments during the insertion, potentially minimizing any trauma caused by the insertion of the implant, ultimately helping preserve residual hearing. This ultimately could lead to improvements in the rates of hearing preservation. Therefore, the current study seeks to investigate: 1) the advantage of using a hearing monitoring system (electrocochleography) monitoring guided CI surgery on hearing preservation rates, 2) determine the benefit that hearing aid/cochlear implant combined hearing provides participants over non-hearing preservation CI (electric-only stimulation from the CI) on measures of speech perception and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Adults, males and females, ages 18 -79 who have a bilateral sensorineural hearing loss with postlingual onset.
3. Minimum of 30 days experience with appropriately fit binaural amplification (standardized National Acoustic Laboratories (NAL) fitting method) verified with real ear measurements within 5 dB SPL of targets.
4. Limited benefit from conventional amplification in the best aided condition as defined by test scores of:

   1. The ear to implanted: Consonant-nucleus-consonant (CNC) words ≤ 60% or AzBio sentences (+10, +5 dB SNR ≤ 60% correct)
   2. Contralateral ear: ≤ 80% on CNC words or AzBio sentences (+10, +5 dB SNR ≤ 80% correct)
5. Low frequency Pure Tone Average (PTA- 125, 250, 500 Hz) ≤ 55 dB HL in the ear to be implanted.
6. Severe to profound mid to high-frequency sensorineural hearing loss (threshold average of 1000, 2000, 3000, and 4000 Hz ≥75 dB HL) in the ear to be implanted.
7. Low frequency PTA ≤ 55 dB HL sloping to moderately severe to profound mid-to high frequency sensorineural hearing loss (threshold average of 1000, 2000, 3000, 4000 Hz ≥ 60 dB) in the contralateral ear.
8. Proficient in English.
9. Undergoing implantation with a current generation CI device from either Cochlear Limited or Advanced Bionics AG.

   1. Cochlear Limited devices include: Nucleus CI612, CI622, CI632, CI624
   2. Advanced Bionics AG devices include: HiFocus SlimJ, Mid-Scala
10. Stated willingness and ability to complete testing and all associated study visits.

Exclusion Criteria:

1. Previous cochlear implantation.
2. Prelingual onset of hearing loss.
3. Abnormal inner ear anatomy on CT imaging.
4. Auditory neuropathy spectrum disorder.
5. Retrocochlear pathology such as a vestibular schwannoma or stroke.
6. Unwillingness or inability to comply with all investigational requirements including the randomization process.
7. Additional medical, or social barriers that would prevent completion of all study requirements.
8. Medical condition contraindicated for surgery.
9. Device selection of Med El CI (per the patient's selection).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Preservation Advantage | 3, 6, 12, 24 months
  Determine the hearing preservation advantage, by measuring low tone audiometry at the 3, 6,12 and 24 month timepoints, in hertz.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Adunka, MD, Principal Investigator — Ohio State University; Amanda Ortmann, PhD, Principal Investigator — Washington University School of Medicine
Locations (5):
- United States (5):
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University Eye and Ear Institute, Columbus, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eggermont JJ. Ups and Downs in 75 Years of Electrocochleography. Front Syst Neurosci. 2017 Jan 24;11:2. doi: 10.3389/fnsys.2017.00002. eCollection 2017. PMID 28174524
- [Background] Gantz BJ, Dunn C, Oleson J, Hansen M, Parkinson A, Turner C. Multicenter clinical trial of the Nucleus Hybrid S8 cochlear implant: Final outcomes. Laryngoscope. 2016 Apr;126(4):962-73. doi: 10.1002/lary.25572. Epub 2016 Jan 12. PMID 26756395
- [Background] Gantz BJ, Hansen MR, Turner CW, Oleson JJ, Reiss LA, Parkinson AJ. Hybrid 10 clinical trial: preliminary results. Audiol Neurootol. 2009;14 Suppl 1(Suppl 1):32-8. doi: 10.1159/000206493. Epub 2009 Apr 22. PMID 19390173
- [Background] Gautschi-Mills K, Khoza-Shangase K, Pillay D. Preservation of residual hearing after cochlear implant surgery: an exploration of residual hearing function in a group of recipients at cochlear implant units. Braz J Otorhinolaryngol. 2019 May-Jun;85(3):310-318. doi: 10.1016/j.bjorl.2018.02.006. Epub 2018 Mar 24. PMID 29631897
- [Background] Gifford RH, Dorman MF, Shallop JK, Sydlowski SA. Evidence for the expansion of adult cochlear implant candidacy. Ear Hear. 2010 Apr;31(2):186-94. doi: 10.1097/AUD.0b013e3181c6b831. PMID 20071994
- [Background] Gstoettner WK, Baumgartner WD, Franz P, Hamzavi J. Cochlear implant deep-insertion surgery. Laryngoscope. 1997 Apr;107(4):544-6. doi: 10.1097/00005537-199704000-00022. No abstract available. PMID 9111389
- [Background] Gstoettner W, Helbig S, Settevendemie C, Baumann U, Wagenblast J, Arnoldner C. A new electrode for residual hearing preservation in cochlear implantation: first clinical results. Acta Otolaryngol. 2009 Apr;129(4):372-9. doi: 10.1080/00016480802552568. PMID 19140036
- [Background] Campbell L, Kaicer A, Sly D, Iseli C, Wei B, Briggs R, O'Leary S. Intraoperative Real-time Cochlear Response Telemetry Predicts Hearing Preservation in Cochlear Implantation. Otol Neurotol. 2016 Apr;37(4):332-8. doi: 10.1097/MAO.0000000000000972. PMID 26859542
- [Background] Herz A, Niedner I, Fraling F, Sommer-Smith J. [Cortical and subcortical reaction potentials after sensory stimulation in wakefull and sleeping cat]. Exp Brain Res. 1966;1(3):249-64. doi: 10.1007/BF00234345. No abstract available. German. PMID 5920552
- [Background] Hodges AV, Schloffman J, Balkany T. Conservation of residual hearing with cochlear implantation. Am J Otol. 1997 Mar;18(2):179-83. PMID 9093674
- [Background] Koka K, Saoji AA, Litvak LM. Electrocochleography in Cochlear Implant Recipients With Residual Hearing: Comparison With Audiometric Thresholds. Ear Hear. 2017 May/Jun;38(3):e161-e167. doi: 10.1097/AUD.0000000000000385. PMID 27879487
- [Background] Lan KK, DeMets DL. Changing frequency of interim analysis in sequential monitoring. Biometrics. 1989 Sep;45(3):1017-20. PMID 2790114
- [Background] Pillsbury HC 3rd, Dillon MT, Buchman CA, Staecker H, Prentiss SM, Ruckenstein MJ, Bigelow DC, Telischi FF, Martinez DM, Runge CL, Friedland DR, Blevins NH, Larky JB, Alexiades G, Kaylie DM, Roland PS, Miyamoto RT, Backous DD, Warren FM, El-Kashlan HK, Slager HK, Reyes C, Racey AI, Adunka OF. Multicenter US Clinical Trial With an Electric-Acoustic Stimulation (EAS) System in Adults: Final Outcomes. Otol Neurotol. 2018 Mar;39(3):299-305. doi: 10.1097/MAO.0000000000001691. PMID 29342054
- [Background] Saoji AA, Patel NS, Carlson ML, Neff BA, Koka K, Tarigoppula VSA, Driscoll CLW. Multi-frequency Electrocochleography Measurements can be Used to Monitor and Optimize Electrode Placement During Cochlear Implant Surgery. Otol Neurotol. 2019 Dec;40(10):1287-1291. doi: 10.1097/MAO.0000000000002406. PMID 31644474
- [Background] Scheperle RA, Tejani VD, Omtvedt JK, Brown CJ, Abbas PJ, Hansen MR, Gantz BJ, Oleson JJ, Ozanne MV. Delayed changes in auditory status in cochlear implant users with preserved acoustic hearing. Hear Res. 2017 Jul;350:45-57. doi: 10.1016/j.heares.2017.04.005. Epub 2017 Apr 12. PMID 28432874
- [Background] Skinner MW, Holden TA, Whiting BR, Voie AH, Brunsden B, Neely JG, Saxon EA, Hullar TE, Finley CC. In vivo estimates of the position of advanced bionics electrode arrays in the human cochlea. Ann Otol Rhinol Laryngol Suppl. 2007 Apr;197:2-24. PMID 17542465